CLINICAL TRIAL: NCT02011581
Title: Diurnal Variability in the Regulation of Beta-cell Function and Insulin Sensitivity in Overweight People
Acronym: 24Hr
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-09110
Record Dates: First submitted 2013-12-09; First posted 2013-12-13 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Overweight
Keywords: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples, adipose tissue samples and muscle samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this research study is to learn more about how our body produces sugar, breaks down fat for fuel, and makes insulin (the major hormone that controls the production of blood sugar and fat breakdown) during a 24-hour day and how body fat and muscle are involved in these processes.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether there are diurnal differences in postprandial beta-cell function and hepatic insulin sensitivity and the factors that influence these metabolic functions, including insulin signaling, adipose tissue and systemic inflammation, nicotinamide phosphoribosyltransferase (NAMPT)-mediated nicotinamide adenine dinucleotide(NAD) biosynthesis, and sirtuin (silent mating type information regulation 2 homolog 1 (SIRT1)) in overweight human subjects.

ELIGIBILITY:
Inclusion Criteria:

* Females
* 18-55 years old
* BMI between 25.0-29.9 kg/m2
* Must be sedentary (regular exercise <1hour/week or <2 times/week

Exclusion Criteria:

* Regular exercise (>1hour/week or >2 times/week)
* Diabetes
* Severe organ dysfunction
* Smokers
* Severe hypertriglyceridemia (>300 mg/dl)
* Medications that may alter the results of the study
* Pregnant
* Breastfeeding

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of female subjects of all races and ethnic groups. Participants will be recruited by reviewing our database of research subjects containing thousands of research study volunteers and by St. Louis metro area postings.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Determine postprandial beta-cell function (insulin secretion) after ingesting breakfast and dinner meals. | 24 hours
  Postprandial pancreatic beta-cell function will be evaluated by using a mixed meal labelled with stable isotope tracers, in conjunction with stable isotope tracer infusion. Metabolic outcomes from the breakfast meal will be compared with values obtained after dinner.
Determine postprandial hepatic insulin sensitivity (suppression of endogenous glucose production) after ingesting breakfast and dinner meals. | 24 hours
  Postprandial pancreatic hepatic insulin sensitivity will be evaluated by using a mixed meal labelled with stable isotope tracers, in conjunction with stable isotope tracer infusion. Metabolic outcomes from the breakfast meal will be compared with values obtained after dinner.

SECONDARY OUTCOMES:
Determine whether there is diurnal variability in muscle insulin signaling | 24 hours
  This muscle samples will be obtained two times (every 12 hours for 24 hours)to assess NAMPT and NAD+ concentrations, SIRT1 activity, and factors involved in insulin signaling.
Determine whether there is diurnal variability in adipose tissue and systemic inflammation. | 24 hours
  Subcutaneous adipose tissue samples will be obtained four times (every 6 hours for 24 hours) to evaluate NAMPT and NAD+ concentrations, SIRT1 activity, and markers of inflammation.
Determine whether there is diurnal variability in NAMPT-mediated NAD+ biosynthesis and SIRT1. | 24 hours
  Blood samples will be obtained at regular intervals for 24 hours to evaluate; 1)plasma free fatty acids (FFA), glucose and insulin concentrations, 2)NAMPT and NAD+ concentrations, 3)SIRT1 activity,and 4)systemic markers of inflammation (C-reactive protein and interleukin (IL) -6).

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Yamaguchi S, Moseley AC, Almeda-Valdes P, Stromsdorfer KL, Franczyk MP, Okunade AL, Patterson BW, Klein S, Yoshino J. Diurnal Variation in PDK4 Expression Is Associated With Plasma Free Fatty Acid Availability in People. J Clin Endocrinol Metab. 2018 Mar 1;103(3):1068-1076. doi: 10.1210/jc.2017-02230. PMID 29294006